CLINICAL TRIAL: NCT05750368
Title: Long-term Outcomes After Epigastric Hernia Repair in Women - a Nationwide Database Study
Acronym: EPI-WOMEN
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Mette Willaume, MD, ph.d., Bispebjerg Hospital
Other Study IDs: women-epigastric
Record Dates: First submitted 2023-02-20; First posted 2023-03-01 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Epigastric Hernia; Women With Epigastric Hernias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women undergoing epigastric hernia repair: all women who have undergone epigastric hernia repair open or laparoscopic in Denmark during af 4-year period from January 1st, 2018, to Dec 31st, 2021.

SUMMARY:
The aim was to evaluate outcomes after epigastric hernia repair in women on a nationwide basis. The primary outcome iss recurrence - secondary outcomes are readmission, operation for complication, risk factors for recurrence, and readmittance.

DETAILED DESCRIPTION:
Aim Outcomes after epigastric hernia repair are rarely reported independently. Furthermore, women have the highest prevalence of epigastric hernia repair in the age of 41-50 years.

The aim of this study was to evaluate long-term outcomes after epigastric hernia repairs in women on a nationwide basis.

Methods Nationwide database cohort study using prospectively recorded data from the Danish Hernia Database from women undergoing elective repair for epigastric hernias, during a 4-year period (2018-2021). A 100% follow-up was obtained by combining intra-operative data with data from the National Civil Register (NRC). The primary outcome was operation for recurrence, secondary outcomes were readmission and operation for complications. We compared open vs. laparoscopic repairs, and subgroup analysis were made for open repairs (sutured vs. mesh).

ELIGIBILITY:
Inclusion Criteria:

* All female patients undergoing elective repair with a laparoscopic or open technique for an epigastric hernia were included.

Exclusion Criteria:

* umbilical or incisional hernias, male patients, recurrent hernia repairs, and hernia repairs performed in relation to other surgical procedures.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — all women undergoing repair
Study Population: all patients undergoing ventral hernia repair in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 3031 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
operation for recurrence | 4 year
  operation for recurrence during the observation period

SECONDARY OUTCOMES:
Readmittance | 90 days
  readmittance within 90 days after repair
operation for complications | 90 days
  90 days operation for complications

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No